CLINICAL TRIAL: NCT07331831
Title: Research on Attitudes, Confidence, and Practical Skills in Performing Cardiopulmonary Resuscitation and Automated External Defibrillation After Completing a Course Based on the European Resuscitation Council Model
Acronym: RACE-CPR
Status: Enrolling by invitation | Type: Observational
Sponsor: First Three Minutes Foundation (Other)
Responsible Party: Principal Investigator, Andrian Georgiev, Researcher, First Three Minutes Foundation
Other Study IDs: FTMF-Res-CPR-001-2025; FTMF-Res-CPR-001-2025 (Other: First Three Minutes Foundation)
Record Dates: First submitted 2025-12-09; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Sudden Cardiac Arrest
Keywords: CPR; AED; Training; Skills; BLS; Attitudes; Confidence
MeSH Terms: conditions — Death, Sudden, Cardiac; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research on attitudes, confidence, and practical skills in performing cardiopulmonary resuscitation and automated external defibrillation after completing a course based on the European Resuscitation Council model

DETAILED DESCRIPTION:
Research on attitudes, confidence, and practical skills in performing cardiopulmonary resuscitation and automated external defibrillation after completing a course based on the European Resuscitation Council model

ELIGIBILITY:
Inclusion Criteria:

* Participation in CPR and AED training course based on ERC standard

Exclusion Criteria:

* No

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical staff, medical students, laypersons.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Trainee CPR and AED practical performance assessed at the end of the course using a 13-item, 4-point Likert scale completed by training instructors. | From beginning to the end of the 4 hour training course
  Practical skills to perform cardio-pulmonary resuscitation and automated defibrillation before and after a training course based on the European Resuscitation Council standard. Assessment of trainee performance (at the end of the course) using a 13-item, 4-point Likert scale completed by training instructors.
Change in self-reported confidence to perform CPR and use an AED assessed using an 11-item, 4-point Likert scale questionnaire before and after training. | From beginning to the end of the 4 hour training course
  Participant confidence to provide cardiopulmonary resuscitation (CPR) and use an automated external defibrillator (AED) is assessed using two standardized self-administered questionnaires completed before and after the training course. Each questionnaire consists of 11 items rated on a 4-point Likert scale. Post-course questionnaire items are rephrased and presented in a different order, while retaining their original meaning. Pre- and post-training scores will be compared to evaluate changes in confidence following the course.
Change in self-reported attitude to perform CPR and use an AED assessed using a 17-item, 4-point Likert scale questionnaire before and after training. | From the beginning to the end of the 4 hour training
  The participant's attitude toward performing cardiopulmonary resuscitation (CPR) and using an automated external defibrillator (AED) is assessed using two standardized self-administered questionnaires, completed before and after the training course. Each questionnaire consists of 17 items rated on a 4-point Likert scale. Post-course questionnaire items are rephrased and presented in a different order, while retaining their original meaning. Pre- and post-training scores will be compared to evaluate changes in attitude following completion of the course.

CONTACTS AND LOCATIONS:
Overall Officials: Mariyana P Manusheva, PhD, Study Director — First Three Minutes Foundation; Andrian Georgiev, PhD, Principal Investigator — First Three Minutes Foundation
Locations (1):
- First Aid School, Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided